CLINICAL TRIAL: NCT01034800
Title: The Neuropsychiatric Evaluation of HIV-Positive and Negative Drug Using Individuals: Study 215
Status: Completed | Type: Observational
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999906300; 06-DA-N300
Record Dates: First submitted 2009-12-16; First posted 2009-12-17 (Estimated); Last update posted 2009-12-17 (Estimated); Status verified 2009-01

CONDITIONS: HIV Infections
Keywords: HIV Positive
MeSH Terms: conditions — HIV Infections; HIV Seropositivity

SUMMARY:
The lack of success in treating substance abuse may be contributed to by a limited understanding of the clinical neurobiology of drug abuse. A better understanding of such deficits might aid in the development of more relevant pharmacological and psychosocial treatment approaches. Thus, the purpose of this study is to test the hypothesis that repetitive illicit drug use may be associated with cortical and subcortical structural abnormalities, vascular abnormalities, as well as neuropsychological decrements. Additionally, a battery of psychological tests are administered to provide information about demographics, drug use, neurocognitive measures, and personality structures....

DETAILED DESCRIPTION:
The lack of success in treating substance abuse may be contributed to by a limited understanding of the clinical neurobiology of drug abuse. A better understanding of such deficits might aid in the development of more relevant pharmacological and psychosocial treatment approaches. Thus, the purpose of this study is to test the hypothesis that repetitive illicit drug use may be associated with cortical and subcortical structural abnormalities, vascular abnormalities, as well as neuropsychological decrements. Additionally, a battery of psychological tests are administered to provide information about demographics, drug use, neurocognitive measures, and personality structures.

ELIGIBILITY:
* Data analysis protocol

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2006-09

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute on Drug Abuse, Biomedical Research Center (BRC), Baltimore, Maryland, United States